CLINICAL TRIAL: NCT02132104
Title: Amnion Graft for Preventing Intrauterine Adhesions Following Hysteroscopic Surgery
Brief Title: Efficiency of Amnion Graft to Prevent Intrauterine Adhesions After Hysteroscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, XUEBING PENG, Associated Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMU-FXH-14-06
Record Dates: First submitted 2014-05-02; First posted 2014-05-07 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Intrauterine Adhesions
Keywords: Intrauterine adhesions; Asherman Syndrome; Amnion graft
MeSH Terms: conditions — Gynatresia | interventions — femoston; Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amnion graft in severe IUA (Experimental): patients, who are with severe IUA, treated by uterine application of amnion membrane + Foley balloon+ hormones (Femoston) following hysteroscopic adhesiolysis.
  Interventions: Procedure: Uterine application of amnion membrane; Device: Foley balloon; Drug: Femoston
- non-amnion graft in severe IUA (Sham Comparator): patients, who are with severe IUA, treated by Foley balloon+ hormones (Femoston) following hysteroscopic adhesiolysis.
  Interventions: Device: Foley balloon; Drug: Femoston

INTERVENTIONS:
Procedure: Uterine application of amnion membrane — Uterine application of amnion membrane following hysteroscopic adhesiolysis.
  Other Names: Human amnion membrane
  Arms: amnion graft in severe IUA
Device: Foley balloon — Uterine application of Foley balloon
Drug: Femoston — Hormones treatment after surgery.
  Other Names: Hormones

SUMMARY:
The purpose of the study is to evaluate whether human amnion graft reduces the reformation of severe intrauterine adhesions (IUA) following hysteroscopic adhesiolysis.

DETAILED DESCRIPTION:
Background

IUA is a consequence of trauma to the endometrium, producing partial or complete obliteration in the uterine cavity and/or the cervical canal, resulting in conditions such as menstrual abnormalities, infertility, and recurrent pregnancy loss. The outcome of hysteroscopic adhesiolysis for IUA is significantly affected by recurrence of intrauterine adhesions. The IUA research should be directed toward reduction of adhesion reformation with a view to improve outcome.

The reformation of intrauterine adhesions appears to be directly related to the severity of the adhesions. It has been reported that the recurrence rate for intrauterine adhesions ranges from 3.1% to 23.5% among all cases of intrauterine adhesions and from 20% to 62.5% in those with severe adhesions.

In this study, considering the high recurrent rate in severe IUA, investigator will focus on severe IUA cases.

Up to now several strategies are commonly employed by various investigators after division of intrauterine adhesions:

1. Physical barriers have been used to promote regeneration of the endometrium and prevention of adhesions. The physical barriers include an intrauterine device (IUD), a Foley catheter, a number of modifications of hyaluronic acid and Auto-cross-linked hyaluronic acid gel.
2. Hormonal treatment has been used to promote regeneration of the endometrium.
3. Antibiotic therapy has been used to prevent infection which is a potent trigger for adhesion formation/reformation.
4. Various medications have been described to increase vascular flow to endometrium, such as asprin, nitroglycerine and sildenafil citrate.

There is published data (Amer et al, 2010), which based on a plot prospective, randomised, comparative study that grafting of either fresh or dried amnion is a promising adjunctive procedure for decreasing recurrence of adhesions and encouraging endometrial regeneration after hysteroscopic lysis of severe intrauterine adhesions. However, the study had a small number of patients, the valid conclusion can not be drawn.

In this study, the aim is to compare the safety and the efficacy of insertion of intrauterine balloon + hormonal treatment with or without grafting amnion to prevent intrauterine adhesion formation/reformation following division of intrauterine adhesions.

Study Design

Patients with severe IUA are enrolled according to the classification of intrauterine adhesion by American Fertility Society.

208 patients with severe IUA were chosen at random and divided equally into those who received amnion graft, following hysteroscopic adhesiolysis (treatment groups) and to those who did not receive the amnion graft (control groups).

Intervention

Following hysteroscopic adhesiolysis, patients will be randomised to have a Foley balloon with or without amnion graft into the uterine cavity. Hormones therapy has been used after surgical treatment both in treatment groups and control groups. A second look and a third look hysteroscopy will be performed about 4 and 12 weeks after the initial operative hysteroscopy. The amount of adhesions, if any, during the initial and reexamine hysteroscopies will be scored.

Power calculation

The investigators' retrospective pilot study data showed that the recurrent rate of severe IUA is around 30% in amnion treatment groups, and around 47.5% in control groups. According to these data, investigators calculated the sample sizes of this study by using Cochran-Mantel-Haenszel test with software PASS 11. Investigators will recruit 104 patients in each group.

Group sample sizes of 104 in group one and 104 in group two achieve 85% power to detect a difference between the group proportions of -0.2000. The group two proportion is 0.5000. The group one proportion is assumed to be 0.5000 under the null hypothesis and 0.3000 under the alternative hypothesis. The test statistic used is the two-sided Z test (unpooled). The significance level of the test was targeted at 0.0500. The significance level actually achieved by this design is not available.

Statistics

Safety and efficacy were evaluated by software NCSS-PASS, using Two Independent Proportions (Non-Null Case) Power Analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for adhesiolysis of intrauterine adhesions
* patients willing to undergo followed hysteroscopy about 4 and 12 weeks after the surgery to assess the reformation of intrauterine adhesions.
* Written, informed consent obtained.

Exclusion Criteria:

* ongoing pregnancy
* Peroperative fever or infections
* Malignancy
* Precious pelvic inflammatory disease
* Uterine fibroid (>3cm size)
* endometriosis
* Contraindications for anesthesia
* Not able to read and/or understand informed consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
safety of intrauterine application of amnion membrane | 3 months
  patients treated by amnion membrane following their hysteroscopic procedure were followed for immediate and late adverse effect: fever, abnormal vaginal discharge, pelvic pain, increased intrauterine adhesion formation upon follow up and changes in menstrual pattern.

SECONDARY OUTCOMES:
efficacy of intrauterine application of amnion graft in reducing adhesion formation following hysteroscopic adhesiolysis. | 3 months
  intrauterine adhesions were assessed and graded according to the American Fertility Society (AFS) score upon hysteroscopy follow up 4 and 12 weeks following initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: TC Li, PhD, Study Director — Hysteroscopic Center, Fu Xing Hospital; Xuebing Peng, MD, Principal Investigator — Hysteroscopic Center, Fu Xing Hospital; Enlan Xia, MD, Study Chair — Hysteroscopic Center, Fu Xing Hospital
Locations (1):
- Fu Xing Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] Amer MI, Abd-El-Maeboud KH, Abdelfatah I, Salama FA, Abdallah AS. Human amnion as a temporary biologic barrier after hysteroscopic lysis of severe intrauterine adhesions: pilot study. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):605-11. doi: 10.1016/j.jmig.2010.03.019. Epub 2010 Jun 23. PMID 20576472
- [Background] Amer MI, Abd-El-Maeboud KH. Amnion graft following hysteroscopic lysis of intrauterine adhesions. J Obstet Gynaecol Res. 2006 Dec;32(6):559-66. doi: 10.1111/j.1447-0756.2006.00454.x. PMID 17100817
- [Background] The American Fertility Society classifications of adnexal adhesions, distal tubal occlusion, tubal occlusion secondary to tubal ligation, tubal pregnancies, mullerian anomalies and intrauterine adhesions. Fertil Steril. 1988 Jun;49(6):944-55. doi: 10.1016/s0015-0282(16)59942-7. No abstract available. PMID 3371491